CLINICAL TRIAL: NCT00002419
Title: A Phase II, 24-Week, Open-Label Study Designed to Evaluate the Safety, Tolerability, and Efficacy of Novel Quadruple-Combination Therapy With Preveon (Adefovir Dipivoxil; Bis-POM PMEA), Abacavir (1592U89), Sustiva (Efavirenz; DMP-266), and Amprenavir (141W94) for the Treatment of HIV-1 Infection in Patients Who Have Failed Previous Protease Inhibitor Treatment
Brief Title: Safety and Effectiveness of Giving Adefovir Dipivoxil Plus Abacavir Plus Efavirenz Plus Amprenavir to HIV-Infected Patients Who Have Failed to Respond to Previous Protease Inhibitor Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Glaxo Wellcome (Industry); Dupont Applied Biosciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 299A; ICC 605
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — abacavir; amprenavir; efavirenz; adefovir dipivoxil

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Efavirenz
Drug: Adefovir dipivoxil

SUMMARY:
The purpose of this study is to see if it is safe and effective to give adefovir dipivoxil plus abacavir (ABC) plus efavirenz (EFV) plus amprenavir (APV) to HIV-infected patients who have failed to respond to previous treatment with protease inhibitors (PIs).

DETAILED DESCRIPTION:
Patients receive a treatment regimen of adefovir dipivoxil, abacavir, efavirenz, and amprenavir for 24 weeks. During the study, patients are evaluated for changes from baseline in plasma HIV-1 RNA levels and lymphocyte subsets and for development of adverse events and toxicities. Patients who experience virologic failure are discontinued from the study. After Week 24, patients with documented virologic response are eligible to continue receiving the study treatment and to attend scheduled follow-up visits.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Had an HIV level of at least 2,000 copies/ml after 6 months of treatment with at least 1 PI other than amprenavir (meaning you failed PI treatment).
* Are at least 13 years old (need consent of parent or guardian if under 18).
* Are able to complete the study.
* Agree to use effective barrier methods of birth control, such as condoms, during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have certain serious medical conditions, including AIDS-related cancers (except Kaposi's sarcoma) that require treatment during the study.
* Have ever taken or are allergic to adefovir dipivoxil, ABC, APV, EFV.
* Are participating in another anti-HIV drug trial during this study.
* Have taken certain medications within 30 days prior to study entry, including medications that affect your immune system.
* Have been diagnosed with hepatitis within the past 30 days.
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.
* Have ever taken NNRTIs.
* Have ever taken ddI or d4T.
* Have received chemotherapy or radiation therapy within 30 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Oaks Med Group, Beverly Hills, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Brown Univ School of Medicine, Providence, Rhode Island
  - Hampton Roads Med Specialists, Hampton, Virginia